CLINICAL TRIAL: NCT00183118
Title: HIV Prevention Partnership in Russian Alcohol Treatment
Brief Title: Russia PREVENT (HIV Prevention Partnership in Russian Alcohol Treatment)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Jeffrey Samet, Professor, General Internal Medicine, Boston Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H23052; R21AA014821 (NIH)
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Alcohol Dependence; Drug Dependence
Keywords: HIV; Russia; Prevention; Behavioral intervention; Alcohol dependence
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Adapted Enhanced-RESPECT (HIV prevention intervention)

SUMMARY:
The purpose of this study is to test an HIV prevention intervention in a Russian substance abuse treatment facility using a randomized trial study design.

DETAILED DESCRIPTION:
A randomized controlled trial of an HIV prevention intervention in a narcology hospital using a stratified randomization design (by gender and substance use diagnosis) will be implemented.

We will conduct a trial among 180 inpatient subjects undergoing treatment at the LRCA. This adapted HIV prevention intervention (adapted Enhanced-RESPECT), Project RESPECT, is a 2-session, one-on-one HIV prevention counseling and testing activity with a trained health educator. By random assignment, half of the subjects will receive the Enhanced-RESPECT intervention, which will include 3 additional booster sessions. And half will receive CDC post-test counseling or standard of care depending on the results of their HIV antibody test. The post-test counseling will follow CDC counseling and testing guidelines. Subjects in the Control group who are not HIV-infected will receive the current standard of care in Russia for non-infected patients; receipt of negative test results by a clinician. HIV pre-test counseling occurs within the first 48 hours of patient arrival at LRCA. CDC post-test counseling guidelines represent a higher standard of care than currently exists within this facility for HIV-infected patients and is equivalent to the standard of care recommended for US HIV testing facilities.

All study participants will be evaluated regarding substance abuse and HIV risk behaviors at baseline and follow-up. Follow up interviews will take place at 3 time points (just before discharge from the hospital and at 3 and 6 months post-randomization). All Intervention participants will receive the basic 2-session adapted RESPECT intervention while inpatients; booster sessions for adapted Enhanced-RESPECT HIV Intervention participants will take place after discharge. Booster sessions will be offered once a month for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years old;
* In-patient at LRCA (i.e., primary diagnosis of alcohol or drug dependence);
* Abstinence from alcohol and other substances of abuse for 4 days;
* Willingness to undergo HIV testing as per standard narcology hospital counseling and testing protocol or known positive HIV serostatus;
* Provision of contact information (e.g., name, home address, telephone number) of two relatives or close friends who can be contacted to share information that may be used to assist with follow-up;
* Stable address within St. Petersburg or districts within 100 kilometers of St. Petersburg; and
* Self-reported unprotected anal or vaginal sex in the last 6 months;

Exclusion Criteria:

* Not fluent in Russian;
* Severe cognitive impairment (Clinically apparent dementia, active psychosis, or severe paranoid disorder) as judged by a narcology hospital clinician and stated in the records;
* Inability to provide informed consent;
* Suspected or diagnosed pulmonary tuberculosis, not receiving treatment;
* Pending legal charges with potential impending incarceration.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2004-10; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
HIV risk behaviors:
risky alcohol use
risky drug use
risky sex behavior

SECONDARY OUTCOMES:
RAB score
Addiction Severity Index (ASI)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey H. Samet, MD, MA, MPH, Study Director — Boston Medical Center; Evgeny Krupitsky, Principal Investigator — Leningrad Regional Center of Addictions Institution: Pavlov State Medical University
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Samet JH, Krupitsky EM, Cheng DM, Raj A, Egorova VY, Levenson S, Meli S, Bridden C, Verbitskaya EV, Kamb ML, Zvartau EE. Mitigating risky sexual behaviors among Russian narcology hospital patients: the PREVENT (Partnership to Reduce the Epidemic Via Engagement in Narcology Treatment) randomized controlled trial. Addiction. 2008 Sep;103(9):1474-83. doi: 10.1111/j.1360-0443.2008.02251.x. Epub 2008 Jul 10. PMID 18636998